CLINICAL TRIAL: NCT06922773
Title: Between the Belly and the Brain: Distorted Gut-brain Crosstalk in Early-life Adversity
Acronym: BellyBrain
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 23275_BELLYBRAIN
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Early Life Adversity; Microbiome, Human; Anxiety Symptoms; Depressive Symptoms; Posttraumatic Stress Symptoms
Keywords: early life adversity; gut microbiome; anxiety symptoms; depressive symptoms; posttraumatic stress symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Faecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Completion of questionnaires; child psychiatric screening; faecal sample analysis — Completion of questionnaires:
  * FFQ (Food Frequency Questionnaire) - completed by child
  * KIDSCREEN-10 - completed by child
  * CRIES-13 (Child Revised Impact of Events Scale) - completed by parents/guardian and child
  * CTES (Childhood Trust Events Survey) - completed by parents/guardian
  * RCADS-25 (Revised Children's Anxiety and Depression Scale) - completed by parents/guardian and child
  Child psychiatric screening using SCID-5-Junior - semi-structured interview conducted with child and parent(s)/guardian
  Faecal sample analysis:
  * Beta-diversity (UniFrac and Bray-Curtis distance index)
  * Firmicutes/Bacteroidetes ratio
  * Abundance of Prevotella, Lactobacillaceae, Bifidobacteriacae and Lachnospiraceae
  * Short-chain fatty acid metabolites

SUMMARY:
The goal of this observational study is to learn about the effects of early-life adversity (ELA) on the composition of children's microbiome and on their psychosocial functioning. The main questions it aims to answer are:

* Do children who have experienced ELA have lower gut microbial diversity and/or an altered gut microbial composition?
* Do these microbiome alterations correlate with adverse neurodevelopmental outcomes, including increased levels of stress, social and/or affective problems?

ELIGIBILITY:
Inclusion Criteria:

* Primary school-aged children (6 to 13 years of age) who have experienced at least one early-life traumatic event, based on the Childhood Trust Events Survey (CTES) questionnaire
* The child and at least one of his/her parents (or guardian) speak Dutch sufficiently well to complete all of the questionnaires and the semi-structured child psychiatric interview (SCID-5-Junior)

Exclusion Criteria:

* any chronic disorders or diseases known to affect the gut micobiome
* inablity to complete questionnaires and/or semi-structured interview because of linguistic and/or cognitive barrier
* congenital or acquired immunodeficiencies
* use of medication(s) that affect gastrointestinal function (e.g., antibiotics) within the last 6 weeks, or laxatives within the last 4 weeks, or probiotic or prebiotic supplements within the last 4 weeks
* current involvement in another clinical or food study

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary school-aged children (6 to 13 years of age) who have been referred to the UZ Brussel child and adolescent psychiatry department
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Global mental wellbeing | Assessment at enrollment
  KIDSCREEN-10 total score
Microbiomial diversity | Assessment based on single stool sample, within 4 weeks after enrollment
  Gut microbiomial beta-diversity, based on UniFrac and Bray-Curtis distance index

SECONDARY OUTCOMES:
Post-traumatic stress symptoms | Assessment at enrollment
  CRIES-13 (Child Revised Impact of Events Scale) total scores, based on parent version and based on child version
Anxiety and depression symptoms | Assessment at enrollment
  RCADS-25 (Revised Children's Anxiety and Depression Scale) total scores, based on parent version and child version
Firmicutes/Bacteroidetes ratio | Assessment based on single stool sample, within 4 weeks after enrollment
  Gut microbiomial Firmicutes/Bacteroidetes ratio
Gut microbiomial composition | Assessment based on single stool sample, within 4 weeks after enrollment
  Gut microbiomial abundance of Prevotella, Lactobacillaceae, Bifidobacteriacae and Lachnospiraceae
Short-chain fatty acid metabolites | Assessment based on single stool sample, within 4 weeks after enrollment
  Gut microbiomial short-chain fatty acid metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium